CLINICAL TRIAL: NCT00251576
Title: A Multicenter, Randomized, Controlled, Double-Blind Trial to Investigate the Clinical Efficacy and Tolerability of Early Treatment With Simvastatin 40 mg Daily for 30 Days, Followed by Simvastatin 80 mg Daily Thereafter in Tirofiban-Treated Acute Coronary Syndrome Patients Who Have Been Randomized to Receive Enoxaparin or Unfractionated Heparin in Conjunction With Aspirin
Brief Title: Aggrastat to Zocor (AtoZ) - the Use of Two Approved Drugs to Treat Patients Who Have Experienced Chest Pain or a Heart Attack (0733-180)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0733-180; 2005_101
Record Dates: First submitted 2005-11-09; First posted 2005-11-10 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Heparin

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: A-Phase: tirofiban; Z-Phase simvastatin
Drug: Duration of Treatment: A-Phase: minimum suggested 48 hours, maximum suggested 108 hours. Z-Phase: 2 years
Drug: Comparator: A-Phase: low molecular weight heparin, unfractionated heparin
Drug: Duration of Treatment: A-Phase: low molecular weight heparin, 2 to 8 days; unfractionated heparin, minium suggested 48 hours, maximum 108 hours
Drug: Duration of Treatment: Z-Phase, 2 years.

SUMMARY:
A-Phase: Evaluating patients with chest pain who are receiving approved drugs, to estimate the effectiveness of one type of blood thinner as compared to another type of blood thinner.

Z-Phase: To evaluate early treatment of patients with long term chest pain (using an approved drug for 30 days, followed by an increased dose of the drug) as compared to patients (treated with diet and 4 months placebo followed by diet and approved drug) in patients who have experienced acute chest pain or heart attack.

ELIGIBILITY:
Inclusion Criteria:

* A-Phase: Chest pain at rest for 10 minutes, EKG changes or elevated cardiac blood work
* Z-Phase: elevated cholesterol , plus at least one risk factor ( > 70 years old, diabetes, history of prior heart or blood vessel disease, chest pain with EKG changes, elevation of cardiac lab work or positive cardiac tests , at least 2 heart vessels blocked [one >= 75% and one >= 50%])

Exclusion Criteria:

* A-Phase: use of some specific cardiac drugs, high risk bleeding, prior blood clotting disorders
* Z-Phase: elevation in certain cardiac blood tests, no significant heart damage at catheterization, planned cardiac surgery or specific cardiac drugs that lower cholesterol levels, within 6 weeks of enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4497 (Actual)
Dates: Start 1999-11-01 (Actual); Primary Completion 2004-03-23 (Actual); Study Completion 2004-03-23 (Actual)

PRIMARY OUTCOMES:
Z-Phase: combined frequency of the following clinical endpoint events: cardiovascular death, MI, readmission for ACS.

SECONDARY OUTCOMES:
Z-Phase: the incidence of the following endpoints, evaluated individually and as a composite: cardiovascular death, MI, readmission for ACS, coronary revascularization due to documented ischemia and non-hemorrhagic stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] de Lemos JA, Blazing MA, Wiviott SD, Brady WE, White HD, Fox KA, Palmisano J, Ramsey KE, Bilheimer DW, Lewis EF, Pfeffer M, Califf RM, Braunwald E; Investigators. Enoxaparin versus unfractionated heparin in patients treated with tirofiban, aspirin and an early conservative initial management strategy: results from the A phase of the A-to-Z trial. Eur Heart J. 2004 Oct;25(19):1688-94. doi: 10.1016/j.ehj.2004.06.028. PMID 15451146
- [Background] de Lemos JA, Blazing MA, Wiviott SD, Lewis EF, Fox KA, White HD, Rouleau JL, Pedersen TR, Gardner LH, Mukherjee R, Ramsey KE, Palmisano J, Bilheimer DW, Pfeffer MA, Califf RM, Braunwald E; Investigators. Early intensive vs a delayed conservative simvastatin strategy in patients with acute coronary syndromes: phase Z of the A to Z trial. JAMA. 2004 Sep 15;292(11):1307-16. doi: 10.1001/jama.292.11.1307. Epub 2004 Aug 30. PMID 15337732
- [Background] Morrow DA, de Lemos JA, Sabatine MS, Wiviott SD, Blazing MA, Shui A, Rifai N, Califf RM, Braunwald E. Clinical relevance of C-reactive protein during follow-up of patients with acute coronary syndromes in the Aggrastat-to-Zocor Trial. Circulation. 2006 Jul 25;114(4):281-8. doi: 10.1161/CIRCULATIONAHA.106.628909. Epub 2006 Jul 17. PMID 16847150
- [Background] Wiviott SD, de Lemos JA, Cannon CP, Blazing M, Murphy SA, McCabe CH, Califf R, Braunwald E. A tale of two trials: a comparison of the post-acute coronary syndrome lipid-lowering trials A to Z and PROVE IT-TIMI 22. Circulation. 2006 Mar 21;113(11):1406-14. doi: 10.1161/CIRCULATIONAHA.105.586347. Epub 2006 Mar 13. PMID 16534008
- [Background] de Lemos JA, Wiviott SD, Murphy SA, Blazing MA, Lewis EF, Califf RM, Pfeffer MA, Braunwald E. Evaluation of the National Cholesterol Education Program Adult Treatment Panel III algorithm for selecting candidates for statin therapy: insights from the A to Z trial. Am J Cardiol. 2006 Sep 15;98(6):739-42. doi: 10.1016/j.amjcard.2006.03.060. Epub 2006 Jul 26. PMID 16950174
- [Result] Morrow DA, de Lemos JA, Blazing MA, Sabatine MS, Murphy SA, Jarolim P, White HD, Fox KA, Califf RM, Braunwald E; Investigators. Prognostic value of serial B-type natriuretic peptide testing during follow-up of patients with unstable coronary artery disease. JAMA. 2005 Dec 14;294(22):2866-71. doi: 10.1001/jama.294.22.2866. PMID 16352794
- [Derived] Morrow DA, Wiviott SD, White HD, Nicolau JC, Bramucci E, Murphy SA, Bonaca MP, Ruff CT, Scirica BM, McCabe CH, Antman EM, Braunwald E. Effect of the novel thienopyridine prasugrel compared with clopidogrel on spontaneous and procedural myocardial infarction in the Trial to Assess Improvement in Therapeutic Outcomes by Optimizing Platelet Inhibition with Prasugrel-Thrombolysis in Myocardial Infarction 38: an application of the classification system from the universal definition of myocardial infarction. Circulation. 2009 Jun 2;119(21):2758-64. doi: 10.1161/CIRCULATIONAHA.108.833665. Epub 2009 May 18. PMID 19451347